CLINICAL TRIAL: NCT03174717
Title: Evaluating an Individualized Music Program Intervention in Long-term Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: David Maggs (Unknown); Jennifer Buckle (Unknown); Veronica Hutchings (Unknown); Kate Lafferty (Unknown); David Tapp (Unknown)
Responsible Party: Principal Investigator, Benjamin Zendel, Canada Research Chair, Assistant Professor, Memorial University of Newfoundland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LTCMusic
Record Dates: First submitted 2017-05-30; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music intervention (Experimental): LTC residents will participate in an individualized music performance with a musician
  Interventions: Behavioral: Music performance

INTERVENTIONS:
Behavioral: Music performance — residents of LTC will learn and perform songs with musicians from the community

SUMMARY:
The goal of this study is to examine the impact of an individualized music program that includes music performance impacts quality of life, PRN drug use and scores on the RAI-MDS for residents of a long-term care facility. The impact of this program on staff at the long-term care facility and musicians performing at the facility will also be assessed.

DETAILED DESCRIPTION:
There is abundant research identifying the value of music in improving quality of life for older adults in residential faculties. This work suggests that there are at least two critical factors that contribute to the success of music-based interventions for older adults: familiarity, and active participation in the production of the music. With these elements in mind, the investigators are proposing to develop a choral singing program comprised of familiar music, introduced to residents at a Long-term care (LTC) facility through individualized engagement with the songs, leading to weekly group participation run by a professional musician at the Bonne Bay (Newfoundland and Labrador, Canada) Long-term Care Facility.

Specific development of the choral program itself will be done through a co-design process involving staff, residents, and care partners during the intervention. In general the intervention will have residents work with professional musicians to select a few songs that the residents will perform with the professional musician at the end of the week. The specific development will determine three crucial issues for the intervention: 1) what music is appropriate for the initiative? 2) what individualized engagements with the songs are appropriate to each resident? 3) what modes of participation in the group events are appropriate to each resident? The key factor with this co-design are that the music and the level of engagement will be tailored to the individual resident.

The program will run over a full quarter in (July, August, September) allowing the investigators to establish meaningful comparisons of secondary, quantitative data already collected at all long-term care facilities on a quarterly basis. This data includes the medication administration (medication administration records: MARS), behavioural episodes in residents with dementia (dementia observational system: DOS), and the resident assessment inventory minimum data set (RAI-MDS). Pre and post intervention data will be assessed for participating residents at the Bonne Bay Long-term care facility. Pre-intervention data will be collected for three years before the intervention to establish an appropriate baseline for the intervention. The impact of the intervention on residents of the unit will also be assessed through qualitative data. Interviews with residents or their care partners will elicit the perceived benefits and challenges to participating in a music intervention program from the participants' point of view. Care-partners will be identified by nursing staff and/or the resident themselves as an individual who regularly helps with day-to-day living needs of the resident. Care partners will only be interviewed when the cognitive abilities of the resident prevent conducting an interview with them. All participants in the study will be de-identified using a code system that allows us to intersect quantitative and qualitative data in pursuit of a more rigorous view of potential impacts. This code system will involve randomly assigning each participant a number. A master database connecting the name and the number will be maintained in a password protected file on a password protected computer in Dr. Zendel's lab. Research staff will use this master database under the supervision of one of the data custodians during the de-identification process.

This intervention will also be studied from the staff perspective. While there are few studies investigating the perceptions of staff in the implementation of music intervention in healthcare settings, those that are published document the importance of considering the staff perspective and the impact of this perspective on the overall success of this form of intervention. A 'pre/post' interview process will engage how the music intervention was perceived by staff, particularly regarding workload, role in the intervention, strengths and challenges of the intervention, and the impact on overall work environment. Gaining an understanding of the staff perspective on the implementation of this intervention will prove invaluable to the overall feasibility of the initiative.

A final layer of inquiry will interview the musicians themselves, exploring a sense of meaning and value gained through participation in the process, distinctions the musicians make between music and music as intervention, how the musician defines and relates to their practice as musicians, what and how that has shifted, what relationship the musician felt emerged between themselves and the residents with whom they worked?

Basic demographic information including age, date of birth and sex will be recorded as part of each interview (residents/care partners, music staff and LTC staff). Demographic information will also be collected from the residents chart.

ELIGIBILITY:
Inclusion Criteria:

* Resident, staff at Bonne Bay LTC, or musician performing at the Bonne Bay LTC

Exclusion Criteria:

* everyone else

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
PRN drug use in LTC residents | 12 weeks
Behavioural assessments | 12 weeks
  RAI-MDS
Experience of LTC residents | 12 weeks
  Qualitative assessment via interview with residents
Experience of LTC staff | 12 weeks
  Qualitative assessment via interview with staff
Experience of Musicians | 12 weeks
  Qualitative assessment via interview with musician

IPD SHARING:
Plan to Share IPD: No